CLINICAL TRIAL: NCT05823831
Title: Social-emotional and Behavioural Problems of Healthcare Workers' Young Children During the Severe Acute Respiratory Syndrome Corona Virus Outbreak: a Case-control Study
Brief Title: Social-emotional and Behavioural Problems of Healthcare Workers During the Outbreak
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, mahmut caner us, M.D., Marmara University
Other Study IDs: 2020.10.2
Record Dates: First submitted 2023-04-20; First posted 2023-04-21 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Emotional Disorder of Childhood
Keywords: Toddlers; Pandemic; Healthcare workers; Socioemotional development; Sleep

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare workers group: Children of healthcare worker mothers were grouped as the Healthcare workers group. Doctors, nurses, and paramedics are considered as healthcare workers.
  Interventions: Diagnostic Test: Brief Infant-Toddler Social and Emotional Assessment (BITSEA) questionnaire; Diagnostic Test: Brief Infant Sleep Questionnaire (BISQ) questionnaire; Diagnostic Test: Multidimensional Scale of Perceived Social Support (MSPSS) questionnaire; Diagnostic Test: Brief Symptom Inventory (BSI) questionnaire
- Non-healthcare worker group: Children of mothers from other occupations were grouped as Non-healthcare workers group
  Interventions: Diagnostic Test: Brief Infant-Toddler Social and Emotional Assessment (BITSEA) questionnaire; Diagnostic Test: Brief Infant Sleep Questionnaire (BISQ) questionnaire; Diagnostic Test: Multidimensional Scale of Perceived Social Support (MSPSS) questionnaire; Diagnostic Test: Brief Symptom Inventory (BSI) questionnaire

INTERVENTIONS:
Diagnostic Test: Brief Infant-Toddler Social and Emotional Assessment (BITSEA) questionnaire — Brief Infant-Toddler Social and Emotional Assessment (BITSEA) questionnaire was used to assess children's social-emotional development.
Diagnostic Test: Brief Infant Sleep Questionnaire (BISQ) questionnaire — A brief Infant Sleep Questionnaire (BISQ) was used to assess children's sleep.
Diagnostic Test: Multidimensional Scale of Perceived Social Support (MSPSS) questionnaire — A Multidimensional Scale of Perceived Social Support (MSPSS) questionnaire was used to evaluate maternal social support.
Diagnostic Test: Brief Symptom Inventory (BSI) questionnaire — A brief Symptom Inventory (BSI) questionnaire was used to evaluate psychological distress.

SUMMARY:
Healthcare worker mothers had to leave their children with their relatives out the fear of contagion and isolated themselves. The investigators aimed to explore the sleep, socioemotional and behavioural problems of children of healthcare workers; assess the psychological distress of mothers and their social support during the Severe Acute Respiratory Syndrome Corona Virus pandemic, and compare them with age-matched children and their mothers from other occupations.

DETAILED DESCRIPTION:
Healthcare worker mothers had to leave their children with their relatives out the fear of contagion and isolated themselves. The investigators aimed to explore the sleep, socioemotional and behavioural problems of children of healthcare workers; assess the psychological distress of mothers and their social support during the Severe Acute Respiratory Syndrome Corona Virus pandemic, and compare them with age-matched children and their mothers from other occupations.

A case-control study design was applied, and a snowball approach was used to enrol volunteered participants aged between 6 to 36 months of age, through a Google survey. The investigators used Brief Infant Sleep Questionnaire and the Brief Infant-Toddler Social and Emotional Assessment questionnaire to assess children's sleep and socioemotional and behavioural problems respectively. A Multidimensional Scale of Perceived Social Support and a Brief Symptom Inventory were used to evaluate the social support and psychological distress of mothers.

ELIGIBILITY:
Inclusion Criteria:

* All women having children aged between 6 to 36 months of age,
* Parental Education above university level,

Exclusion Criteria:

* Out of age range,
* Parental Education below university level
* Didn't read the informed consent form and tick the mandatory consent box

Ages: 6 Months to 36 Months | Sex: All
Age Groups: Child
Study Population: All women having children aged between 6 to 36 months of age
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Social-emotional and behavioural problems of healthcare workers children | Baseline
  The study was planned based on the hypothesis that children of healthcare workers experienced more socioemotional and behavioural problems than children of mothers from other occupations during the Severe Acute Respiratory Syndrome Corona Virus pandemic. The investigators aimed to explore Social-emotional and behavioural problems of healthcare workers by using Brief Infant-Toddler Social and Emotional Assessment (BITSEA) questionnaire, and compare them with age-matched peers and their mothers from other occupations.

SECONDARY OUTCOMES:
Sleep problems of healthcare workers children | Baseline
  The investigators aimed to explore Sleep problems of healthcare workers by using Brief Infant Sleep Questionnaire (BISQ) questionnaire, and compare them with age-matched peers and their mothers from other occupations.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Caner Us, M.D., Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Diver S, Buccheri N, Ohri C. The value of healthcare worker support strategies to enhance wellbeing and optimise patient care. Future Healthc J. 2021 Mar;8(1):e60-e66. doi: 10.7861/fhj.2020-0176. PMID 33791478
- [Background] Halley MC, Mathews KS, Diamond LC, Linos E, Sarkar U, Mangurian C, Sabry H, Goyal MK, Olazo K, Miller EG, Jagsi R, Linos E. The Intersection of Work and Home Challenges Faced by Physician Mothers During the Coronavirus Disease 2019 Pandemic: A Mixed-Methods Analysis. J Womens Health (Larchmt). 2021 Apr;30(4):514-524. doi: 10.1089/jwh.2020.8964. Epub 2021 Mar 23. PMID 33761277
- [Background] Skokauskas N, Leventhal B, Cardeli EL, Belfer M, Kaasboll J, Cohen J. Supporting children of healthcare workers during the COVID-19 pandemic. Eur Child Adolesc Psychiatry. 2022 Jan;31(1):203-204. doi: 10.1007/s00787-020-01604-6. Epub 2020 Jul 18. No abstract available. PMID 32683490
- [Background] Prime H, Wade M, Browne DT. Risk and resilience in family well-being during the COVID-19 pandemic. Am Psychol. 2020 Jul-Aug;75(5):631-643. doi: 10.1037/amp0000660. Epub 2020 May 21. PMID 32437181
- [Background] Zhang J, Deng X, Liu H, Xu X, Fang R. Evaluation of the mental health status of community healthcare workers during the COVID-19 outbreak. Medicine (Baltimore). 2021 Feb 12;100(6):e24739. doi: 10.1097/MD.0000000000024739. PMID 33578622